CLINICAL TRIAL: NCT02118805
Title: Quantitative Ultrasonography and Electrical Impedance Myography: Speech and Swallowing Technologies for Use in Neurological Disorders
Brief Title: Innovative Measures of Speech and Swallowing Dysfunction in Neurological Disorders
Acronym: QUESST
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Seward Rutkove, Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2013P000204
Record Dates: First submitted 2014-04-08; First posted 2014-04-21 (Estimated); Last update posted 2024-04-16 (Actual); Status verified 2023-04

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Myasthenia Gravis; Myopathies; Stroke; Parkinson's Disease
Keywords: ALS; Myasthenia Gravis; Myopathy; Stroke; Parkinson's Disease; Bulbar; Orofacial; Ultrasound; Electrical Impedance Myography
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Myasthenia Gravis; Muscular Diseases; Stroke; Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Patients with ALS: No intervention is used in this study. The health of muscle is monitored over time.
- Patients with Myasthenia Gravis: No intervention is used in this study. The health of muscle is monitored over time.
- Patients with Muscle Disease: No intervention is used in this study. The health of muscle is monitored over time.
- Patients with Stroke: No intervention is used in this study. The health of muscle is monitored over time.
- Patients with Parkinson's Disease: No intervention is used in this study. The health of muscle is monitored over time.
- Healthy Volunteers: No intervention is used in this study. The health of muscle is monitored over time.

SUMMARY:
This study is evaluating the use of two painless, non-invasive technologies in the assessment of muscle health over time in both healthy volunteers and patients who have diseases that affect the nervous system.

DETAILED DESCRIPTION:
Speech and swallowing abnormalities are important symptoms associated with disorders of the central nervous system, motor neuron disease (such as amyotrophic lateral sclerosis), myasthenia gravis, and primary muscle conditions. In addition to characterizing the evolution in muscle architecture that could underlie associated orofacial weakness, identifying new ways to measure these abnormalities is critical to the development and testing of novel treatment approaches. As painless, non-invasive, portable technologies, quantitative ultrasonography (QUS) and electrical impedance myography (EIM) could meet the need for objective measures of speech and swallowing dysfunction.

In QUS, acoustic energy is applied to a muscle of interest; the resultant pictorial data are translated into a single value that reflects the health of the imaged muscle. Similarly, in EIM, a high-frequency, low-intensity alternating electrical current is applied to individual muscles, and the resulting voltages measured. Impedance values reflect changes in muscle architecture, including fiber atrophy, inflammation, and the replacement of muscle with fat or connective tissue. Both of these user-friendly methods can provide sensitive indicators of neuromuscular disease status when applied to the limbs. Although they have also been used to evaluate orofacial muscles in healthy volunteers and patients with primary muscle disorders, they have not yet been systematically studied in patients with a range of neurological conditions.

When applied to muscles of the face and tongue, such tools could 1. Improve accuracy of early diagnosis; 2. Allow monitoring of speech and swallowing dysfunction over time; 3. Help individualize care; and 4. Serve as biomarkers in clinical trials. We propose that QUS and EIM will provide convenient, reliable, clinically meaningful surrogate markers of orofacial dysfunction in a variety of neurologic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Established, or clinically probable, neurologic diagnosis with at least the potential for associated bulbar dysfunction
* Age 20-90 years

Exclusion Criteria:

* History or presence of a medical condition that substantially impacts bulbar function
* Age under 20 or over 90 years

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited principally from the BIDMC outpatient clinics and inpatient ward service. Healthy volunteers will be recruited through online advertising.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Health over 18 months by Standard Ultrasound | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Selected muscles of the face, limbs, trunk, and tongue will be visualized with painless, non-invasive ultrasound; this measure will be performed in healthy volunteers and participants with neurological conditions

SECONDARY OUTCOMES:
Change in Score on the Sydney Swallow Questionnaire (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants with neurological conditions will answer questions about swallowing
Change in Number of Seconds It takes to Repeat Individual Words Ten Times (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants with neurological conditions will be asked to repeat "pepper" and "ticker" ten times as quickly as possible
Change in Number of Seconds It Takes to Swallow of 3 ounces of Water (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants with neurological conditions will be asked to perform this task if safe
Change in Score on the Amyotrophic Lateral Sclerosis Rating Scale - Revised (ALSFRS-R) (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants who have been diagnosed with ALS will answer questions about function, including speech and swallowing
Change in Score on the Quantitative Myasthenia Gravis Scale (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants who have been diagnosed with Myasthenia Gravis will be asked to perform certain tasks, such as raising the arm, and the findings will be scored by a research team member
Change in Score on the United Parkinson's Disease Rating Scale (UPDRS) (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants who have been diagnosed with Parkinson's Disease will be asked questions about function, including speech and swallowing
Change in Muscle Health by Standard Concentric Needle Electromyography (EMG) (over 18 months) | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Participants who have been diagnosed with ALS will be asked if they are willing to participate in standard needle EMG of selected muscles of the face and tongue
Change in Muscle Health by Specialized Electrical Impedance Arrays | Baseline, Month 3, Month 6, Month 9, Month 12, Month 15, and Month 18
  Selected muscles of the face, limbs, trunk, and tongue will be measured using painless, specialized electrode arrays; this measure will be performed in healthy volunteers and participants with neurological conditions

CONTACTS AND LOCATIONS:
Overall Officials: Seward Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States